CLINICAL TRIAL: NCT01319123
Title: Clinical Study to Comparatively Evaluate the Impact of Drawtex Wound Dressing Against Wound Bioburden in Moderately to Highly Exuding Venous Leg Ulcers
Brief Title: Evaluate the Impact of Drawtex in Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Regional Wound Care Center (Other)
Collaborators: Beier Drawtex Healthcare, (PTY). Ltd (Unknown)
Responsible Party: Principal Investigator, Randall Wolcott, Principal Investigator, Southwest Regional Wound Care Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56-RW-019
Record Dates: First submitted 2011-03-10; First posted 2011-03-21 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Moderatley to Highly Exuding Venous Leg Ulcers
Keywords: dressing for venous leg ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- wound dressing (Other): The dressing is indicated for moderately to heavily exuding wounds such as venous leg ulcers.
  Interventions: Device: Drawtex dressing

INTERVENTIONS:
Device: Drawtex dressing — The dressing is indicated for moderately to heavily exuding wounds such as venous leg ulcers
  Other Names: Beier Drawtex

SUMMARY:
This is a clinical study to comparatively evaluate the impact of Drawtex wound dressing against wound bioburden in moderately to highly exuding venous leg ulcers.

DETAILED DESCRIPTION:
Each subject is expected to participate in this study for a period of four weeks or until reepithelialization, whichever occurs first. Subjects may participate for an additional period of four weeks or until reepithelialization, whichever occurs first: this it to be decided by the investigator and will be determined by the accessibility of the patient (physical location) and the suitability of the wound to further treatment. The maximum time period for the study is 8 weeks. The minimum time frame is at least 4 week, or until reepithelialization occurs.

ELIGIBILITY:
Inclusion Criteria:

* Subject > 18 years.
* Subject is attending weekly office visits at SW Wound Care Center as an out-patient.
* Subject has a moderately to highly exudative venous leg ulcer that would be indicated for treatment with Drawtex
* Subject or is informed about the trial, understands its nature of the study and provides written informed consent prior to study enrollment.
* Subject is willing and able to comply with all specified care and visit requirements

Exclusion Criteria:

* Subject has a lesion that does not meet the inclusion criteria.
* Subject refuses to participate in the study.
* Subject already participates in the this study with one wound (only one wound per subject is allowed)
* Subject has known sensitivity to the trial product or any of its compounds.
* Subject is expected to be non-compliant.
* Subject's lesion is a primary skin cancer.
* Subject's lesion is the manifestation of a metastasis.
* Subject is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To investigate the impact of Drawtex on wound surface bioburden. | 2 years
  The dressing is indicated for moderately to heavily exuding wounds such as venous leg ulcers.• The safety of Drawtex will be measured by the number and type of any adverse events. Patient's tolerance and acceptance of the different dressings

SECONDARY OUTCOMES:
Tolerance | 2 years
  To further investigate whether Drawtex
  * Will have an overall benefit on the wound healing process.
  * Patient's tolerance and acceptance of the dressings. The overall effect on wound healing, as expressed by percentages of necrosis, slough, granulation and/or epithelium at the wound surface.
  * Condition of periwound skin
  * Mobility restrictions, related to the dressing
  * The number of dressings per dressing change, the number of dressing changes and the amount of nursing time involved

CONTACTS AND LOCATIONS:
Overall Officials: Randall D Wolcott, M.D., Principal Investigator — Southwest Regional Wound Care
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States